CLINICAL TRIAL: NCT02820545
Title: Patient's Perception of Hospital Safety: Measure of the Patients' Perception and Correlation With Patient Safety Strategies in the Surgical Care Units
Brief Title: Patient's Perception of Hospital Safety
Acronym: PERSEPOLIS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14_0452
Record Dates: First submitted 2016-06-13; First posted 2016-07-01 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Patient Safety in Surgical Care Units
Keywords: patient safety culture; hospital; patient perception; healthcare professional perception; sociological; qualitative; questionnaire construct; psychometrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sociological interview: Patients will take a sociological interview with a sociologist during their hospital stay
  Interventions: Other: Sociological interview
- Self-administrated questionnaire: Patients will take a self-administrated questionnaire at the end of their hospital stay and one week after they left hospital
  Interventions: Other: Self-administrated questionnaire

INTERVENTIONS:
Other: Sociological interview — A sociological interview will be performed with each patient by a sociologist, during their hospital stay
  Groups: Sociological interview
Other: Self-administrated questionnaire — Self-administrated questionnaire will be performed by patients themselves at the end of hospital stay and one week after they left hospital
  Groups: Self-administrated questionnaire

SUMMARY:
The study aims to construct and validate a self-administrated questionnaire to assess the patients' perception of patient safety in surgical care units. The originality of the study is to perform sociological interviews of hospitalized patients to assess their own perception on the safety of their care and to create corresponding items which will be included in a new questionnaire. In a second step, patients' perception of patient safety will be assessed in numerous surgical care units in France, in order to analyze the psychometric properties of the questionnaire and consequently to validate the questionnaire. The patients' perception will be compared to the healthcare professionals' perception on patient safety and to the patient safety strategies in place in the care units.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in a surgical care unit for at least 1 night stay
* Patient hospitalized for a scheduled surgery
* French speaking patient

Exclusion Criteria:

* Ambulatory surgery
* Hospitalization in emergency
* Unable to answer a survey
* Patient transfer from another unit of the same hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in surgical care units
Sampling Method: Non-Probability Sample
Enrollment: 1277 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Patient's perception of patient safety in hospital measured by sociological interviews (qualitative outcome) | During patient's hospital stay, up to 2 weeks
  This qualitative outcome is measured by sociological interviews of hospitalized patients to construct a new questionnaire. Sociological interviews will be analyzed to identify items and dimensions of the patient's perception to introduce in the questionnaire.

SECONDARY OUTCOMES:
Care safety perception score | 7 days after patient left hospital
  This score is measured by patient himself thanks to the self-administrated questionnaire
Care safety perception score | The day patient leave hospital, up to 2 weeks
  This score is measured by patient himself thanks to the self-administrated questionnaire
Patient Safety Strategies (PSS) score | During patient's hospital stay, up to 2 weeks
  The PSS questionnaire is completed for each patient by health care professionals

CONTACTS AND LOCATIONS:
Overall Officials: Pauline OCCELLI, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Pole Information Médicale Evaluation Recherche, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Occelli P, Mougeot F, Robelet M, Buchet-Poyau K, Touzet S, Michel P. Feelings of Trust and of Safety Are Related Facets of the Patient's Experience in Surgery: A Descriptive Qualitative Study in 80 Patients. J Patient Saf. 2022 Aug 1;18(5):415-420. doi: 10.1097/PTS.0000000000000950. Epub 2021 Dec 17. PMID 35948291